CLINICAL TRIAL: NCT02978209
Title: Double Blinded Randomized Clinical Study of Carbamide as Moisturizer in Ichthyosis Vulgaris
Brief Title: Comparison of Different Concentrations of Carbamide as Moisturizers in Ichthyosis Vulgaris
Acronym: Urea-IV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UFKOPAUH201601
Record Dates: First submitted 2016-11-08; First posted 2016-11-30 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-02

CONDITIONS: Ichthyosis Vulgaris
MeSH Terms: conditions — Ichthyosis Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Only moisturizer, no carbamide (No Intervention): 20 patients with Ichthyosis Vulgaris at age 0-80 years old. One body half
- Moisturizer + 7,5 % carbamide (Active Comparator): 20 patients with Ichthyosis Vulgaris at age 0-80 years old. Other body half
  Interventions: Device: 7.5 %

INTERVENTIONS:
Device: 7.5 % — Patient untreated with moisturizers for 1-2 weeks will start applying moisturizers containing urea at concentration 0 % on one half of the body twice a day while applying the same moisturizer with 7.5 % urea on the other half of the body in the same quantity at the same frequence
  Other Names: Carbamide = Urea
  Arms: Moisturizer + 7,5 % carbamide

SUMMARY:
A randomized double blinded clinical trial will be conducted comparing the effect of two simple basic moisturizers only different in the concentration of carbamide (urea). The concentrations of carbamide will be tested are 0 and 7.5, respectively. The study will be conducted as a split-body-study and will contain two arms randomized to comparing 0 and 7.5 % carbamide, respectively. Approximately 20 patients with at least clinically verified Ichthyosis Vulgaris will be enrolled to each study arm. The effect of the moisturizers will be assessed by clinical examination (score), patients assesment of effect and measurement of transepidermal water loss (TEWL) and other skin parameters.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Ichthyosis Vulgaris

Exclusion Criteria:

* All other forms of Ichthyosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Skin dryness | 2-8 weeks
  Transepidermal water loss ('TEWL) (g/m2/h)

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Koppelhus, MD, PhD, Principal Investigator — Associate professsor
Locations (1):
- Department of Dermatology, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Dorf ILH, Lunen MS, Koppelhus U. Effect of topical treatment with 7.5% urea in Ichthyosis Vulgaris: A randomized, controlled, double blinded, split body study evaluating the effect of urea cream compared to the vehicle (moisturizing) cream. Skin Health Dis. 2021 Sep 14;1(4):e65. doi: 10.1002/ski2.65. eCollection 2021 Dec. PMID 35663767